Version No: 14

Version Date: November 14, 2023

Clinical impact of a volumetric image method for confirming tumor coverage with

Ablation on patients with malignant Liver Lesions

(COVER-ALL)

Principal Investigator: Bruno C. Odisio MD

Co-Investigators: Kristy K. Brock, PhD, Jean-Nicolas Vauthey, MD, Sanjay Gupta,

MD, Scott Kopetz, MD,

Collaborators: HyunSeon Kang, MD, Veronica Cox, MD, Ahmed Kaseb, MD, Imad

shureiqu, MD, Kanwal Raghav, MD, Michael Overman, MD, Joshua Kuban, MD,

Kamran Ahrar, MD, Ching-Wei Tzeng, MD, Yun Shin Chun, MD, Bryan Fellman,

Hop Tran Cao, MD, Milind Javle, MD, Van K Morris, MD, Timothy Newhook, MD,

Zeyad Metwalli, MD, Ketan Yogesh Shah, MD, Milan Patel, MD

Statistician: Bryan Fellman

Outside collaborator: Joe E Ensor PhD - Houston Methodist Cancer Center,

Houston Methodist Research Institute, jeensor@houstonmethodist.org, 6670

Bertner Ave, Houston, 77030


| | l impact of a volumetric image method for confirming tumor coverage with Ablatio | • |
|---|---|---|
| with m | nalignant Liver Lesions | 1 |
| (COVE | R-ALL) | 1 |
| Princip | oal Investigator: Bruno C. Odisio MD | 1 |
| Co-Inve | estigators: Kristy K. Brock, PhD, Jean-Nicolas Vauthey, MD, Sanjay Gupta, MD, Scot | t Kopetz, MD, 1 |
| Raghav<br>Wei Tz | orators: HyunSeon Kang, MD, Veronica Cox, MD, Ahmed Kaseb, MD, Imad shureiqu<br>v, MD, Michael Overman, MD, Joshua Kuban, MD, Steven Y. Huang MD, Kamran Ah<br>eng, MD, Yun Shin Chun, MD, Bryan Fellman, Hop Tran Cao, MD, Milind Javle, MD,<br>mothy Newhook, MD, Zeyad Metwalli, MD, Ketan Yogesh Shah, MD | rar, MD, Ching-<br>Van K Morris, |
| Statisti | ician: Bryan Fellman | 1 |
| | e collaborator: Joe E Ensor PhD - Houston Methodist Cancer Center, Houston Meth te, jeensor@houstonmethodist.org, 6670 Bertner Ave, Houston, 77030 | |
| List of A | Abbreviations | 3 |
| OBJECT | TIVES | 4 |
| 1.1 | Primary Objective | 4 |
| 1.2 | Secondary Objectives | 4 |
| BACKG | GROUND | 4 |
| 1.3 | Rationale | 4 |
| 1.4 | Clinical Impact | 6 |
| 1.5 | Mechanism | 9 |
| ELIGIBI | ILITY | 12 |
| 1.6 | Inclusion Criteria | 12 |
| 1.7 | Exclusion Criteria | 13 |
| NUMB | ER OF PARTICIPANTS | 13 |
| 1.8 | Method | 14 |
| 1.9 | Collecting Time Points | 20 |
| PROCE | DURE TO OBTAIN CONSENT | 20 |
| PATIEN | NT INFORMATION AND CONFIDENTIALITY PLAN | 20 |
| STATIS <sup>*</sup> | TICAL CONSIDERATIONS | 21 |
| PROTO | OCOL MONITORING PLAN | 24 |
| DATA ( | COLLECTION PLAN | 25 |


| REFERENCES | 27 |
|-------------------------------|----|
| QUESTIONNAIRES | 30 |
| QUALITY OF LIFE QUESTTIONAIRE | 32 |

## **List of Abbreviations**

ASA: American society of anesthesiologists

CECT: contrast-enhanced computed tomography

CLM: colorectal liver metastasis

CT: computed tomography

DIR: deformable imaging registration

DTA: distance to agreement

ECOG: eastern cooperative oncology group classification

FEA: finite element analysis

INR: international normalized ratio

LTP: local tumor progression

LTPF: local tumor progression-free survival

MAM: minimal ablation margins

MR: magnetic resonance

MW: microwave ablation

OS: overall survival

PTA: percutaneous ablation

QOL: quality of life

RFA: radiofrequency ablation

TRE: target registration error


**OBJECTIVES** 

1.1 Primary Objective

To evaluate if the intra-procedure feedback of a biomechanical deformable

registration volumetric image method during percutaneous ablation will increase the

minimal ablation margins on a three-dimensional computed tomography-generated

analysis.

1.2 Secondary Objectives

1. To assess whether applying the proposed method during percutaneous ablation

improves local tumor progression-free survival (LTPFS) rates;

2. Evaluate impact of software use on procedure workflow;

3. Impact of software use on complication rates, quality of life, liver function;

4. Evaluate oncological outcomes (intra-hepatic and overall progression-free survivals,

and overall survival)

**BACKGROUND** 

1.3 Rationale

Primary liver cancer is the second leading cause of death worldwide with an

estimated 788.000 related-deaths in 2015. The global burden of primary liver cancer can

also be demonstrated by the impact on disability-adjusted life-years, which was estimated


in 20.578.000 in 2015. In addition to primary liver cancer, approximately two-thirds of all the 774.000 colorectal cancer-related deaths - the third most common cause of cancer-related death worldwide and the most common cause of metastatic liver cancer - are attributed to the presence of colorectal liver metastasis (CLM). Collectively, primary and secondary liver cancers are responsible for over 1 million deaths per year worldwide. Moreover, it is expected an increase on the incidence on both primary and secondary liver cancers in the next decades owing to population growth and aging. Therefore,

effective therapies for the treatment of primary and secondary liver cancers are needed.

Among the curative treatments available for primary liver cancer, surgical resection (or liver transplantation) and ablation are both considered the standard of care on patients with very early and early stage accordingly to the Barcelona Clinic Liver Cancer staging and treatment strategy (1). Contrarily, for secondary liver cancers such as colorectal cancer liver metastasis, surgical resection is still considered the modality of choice. Unfortunately, only 20% of the patients with colorectal liver metastasis are considered surgical candidates (2), with percutaneous thermal ablation used as an acceptable alternative for the remaining of the non-surgical candidates (3), highlighting the importance of this therapy as a therapeutic option. Moreover, results of prospective phase II randomized clinical trial demonstrated improved overall survival rates among patients treated with a combination of percutaneous liver ablation and systemic chemotherapy for CLM when compared to patients treated with systemic chemotherapy alone (4).

Currently, several ablation modalities are available for clinical use. Among those, radiofrequency ablation (RFA) and microwave (MW) coagulation are the most commonly


utilized. Such modalities have fundamental differences in the way tumor destruction is

obtained. RFA promotes tumor destruction by the delivery of an alternating electrical

current within the tumor resulting in frictional heat and movement of electrons within the

lesion and surrounding tissues, whereas MW promotes tissue heating by causing polar

water molecules to continuously realign with an oscillating electromagnetical field that

emanates from the microwave antenna. Both technologies produces tissue friction and

heat induces cellular destruction via coagulative necrosis. More recently, MW has been

used more frequently in clinical practice given its advantages in achieving higher ablation

temperatures and larger ablation zones. Nevertheless, when compared to RFA, MW is

associated with a lower level of predictability between the desired ablation zone planned

and the actual ablation zone achieved. Such discrepancy might affect both the safety of

the procedure (i.e. larger unanticipated ablation zones with damage of critical structures

adjacent to the ablated tumors) as well the oncological outcome of it (i.e. smaller ablation

zone not encompassing the entire tumor volume). Moreover, tissue volumetric loss are

more prominent with MW coagulation when compared to RFA, which limits the ability of

the operator to ascertain with confidence adequate tumor coverage. Therefore, tailored

high-precision image-guidance during ablation is critical for reducing procedure-

associated complications and achieve optimal outcomes.

1.4 Clinical Impact

Among the local therapies utilized for liver cancers, percutaneous thermal ablation

has become a widely utilized option for patients not eligible for surgery, with most recent

series demonstrating similar 5-year overall survival rates between surgery and ablation


(5-7). This highlights the efficacy of this treatment modality on prolonging OS in patients with liver cancers (4).

In order to achieve optimal results with ablation, low rates of local recurrence (also known as local tumor progression [LTP]) at the treated tumors should be obtained. More recently, results of a prospective randomized phase II trial demonstrated that patients with CLM treated liver ablation in association with systemic chemotherapy had significantly longer overall survival rates (OS) when compared to patients treated only with systemic chemotherapy (4), emphasizing the role of aggressive local treatment on prolonging OS in patients with unresectable CLM. In an effort to improve local disease control and oncologic outcomes after liver ablation, several factors have been studied (15-19). Among the known factors associated with improved local tumor control with ablation, lesion diameter < 3 cm, number and location of tumors, and minimal ablation margins achieved around the target tumor(s) are widely recognized as critical variables, with the latter being the only one passive for modification during treatment delivery. Moreover, it has been recently described that biological factors such as the RAS mutational status are also prognostic indicators for local recurrence and survival in patients undergoing ablation of CLM and have prompted recommendations for wider ablation margins in patients with RAS-mutated tumors (8, 20), suggesting that the minimal ablation margin acceptable for optimal disease control needs to be tailored to distinct tumor subtypes.

In order to provide adequate ablation margins, several elements are important: firstly, it is critical to have optimal definition of the tumor extent on intra-procedural CT


image; secondly, confirmation of precise probe placement in relation to the tumor is

needed intra-procedurally; thirdly, the volumetric loss and peri-tumoral tissue

inflammation promoted by the ablation limits the ability to evaluate with confidence the

ablation margin intra-procedurally, therefore requiring a magnetic resonance (MR) or

computed tomography (CT) study to be performed within 1-2 months following ablation

procedure, a long period to evaluate the primary efficacy of this modality. Taking all

together, those factors points to the need of having improved intra-procedurally imaging

assessment of patients undergoing percutaneous ablation.

Currently, there are no commercially available tools that provide a robust and

accurate method for tumor mapping and ablation confirmation that takes in consideration

the biomechanical conformational changes promoted by this therapy. We hypothesize

that local tumor control following percutaneous ablation of liver cancers will be

significantly improved with the application of a dedicated anatomical linear elastic

biomechanical model for treatment guidance and efficacy assessment by enabling the

operator to accurately identify the tumor for ablation probe placement and assess intra-

procedurally the minimal ablation margins, therefore increasing efficacy of percutaneous

ablation therapy, ultimately improving liver progression-free survival rates.

Our preliminary data shows that our biomechanical model can accurately map the

tumor, defined on pre-treatment computed tomography (CT) imaging, onto an intra-

procedural CT image and is insensitive to imaging artifacts associated with ablation

probe. We hypothesize that our innovative approach to modeling the tissue changes

related to the ablation procedure will enable intra-procedure monitoring of the ablation


margin relative to the tumor. In addition, the combination of these technologies will provide further detailed information on the relationship between progression-free survival local tumor progression-free survival (LTPFS) and the ablation margins achieved.

#### 1.5 Mechanism

A multi-organ finite element model (FEM)based deformable image registration (DIR)

Contoured Reference Surface Planning CT Mesh Assign material 1.97 properties 1.48 Apply boundary conditions to drive Test Surface -0.49CBCT – contours surface correlation of generated Mesh organs Use Finite Element Analysis to yield DVF

method (Morfeus) has

been developed in a

Figure 1. Morfeus schematic. Contours from reference volume (planning CT) and test volume (generated semi-automatically) are matched by Finite Element analysis

previously funded R01 and extensively validated on several sites including head and neck, lung, liver, stomach, esophagus, pancreas, prostate, rectum, cervix, and extremity sarcoma (8-29). A commercially available FEM pre and post processes (HyperMesh, Altair Engineering, Troy, MI) and a Finite Element Analysis (FEA) software package (ABAQUS, ABAQUS Inc, Pawtucket, RI) are utilized for model creation and analysis. Morfeus, is briefly described below, illustrated in Figure 1, and described in detail in the referenced publications: Briefly, manual contouring of regions of interest are generated and converted to a 2D surface mesh (clouds of nodes, connected to form elements). The number of elements can be reduced, leading to increase in efficiency, by combining elements and smoothing regions of high frequency.


This surface mesh is a shell from which a 3D volume mesh is created, consisting of tetrahedral elements. Multi-organ models are created by constructing surface interfaces between neighboring region of interest meshes to govern their interaction. Boundary conditions, or loads applied to the FEM (e.g. force, moment, constraint, or pressure), provide a relationship between the initial and secondary representation of the mesh. Preliminary investigations focused on the use of applied constraints, or set displacements, assigned to a subset of elements in the model, determined by projecting the nodes on the surface of one region of interest onto a surface representation of the same region of interest constructed from another imaging session. Finite Element Analysis (FEA) determines the results of the boundary conditions for all nodes in the model. In summary, the method does not explicitly use intensity information in the registration, only for the manual delineation of regions of interest, the registration process is identical for images of the same or different modalities, the registration is driven by the alignment of a subset of the region of interest surfaces using a guided surface projection method, and the full deformation map (i.e. points in space with defined displacements), relating two images, is calculated using biomechanical models and solving the constitutive equations using FEA.

This algorithm was licensed to RaySearch Laboratories (Stockholm, Sweden) for integration into their radiation therapy treatment planning system RayStation. The algorithm was extensively validated to confirm that the integration was performing with the same accuracy as the in-house developed system. Overall, the mean distance to agreement (DTA) was ≤ 1.0 mm for controlling structures (i.e. the liver) and 1.0–3.5 mm


for implicitly deformed structures (i.e. the kidneys) on average. Target registration error

(TRE) ranged from 2.0 mm on prostate MR to 5.1 mm on lung MR on average, within 0.1

mm or lower than the image voxel sizes. Accuracy was not overly sensitive to changes in

the material properties or variability in structure segmentations, as changing these inputs

affected DTA and TRE by ≤ 0.8 mm. Maximum DTA > 5 mm occurred for 88% of the

structures evaluated although these were within the inherent segmentation uncertainty

for 82% of structures. Differences in accuracy between the commercial and in-house

research implementations were  $\leq 0.5$  mm for mean DTA and  $\leq 0.7$  mm for mean TRE.

Deformable image registration for multi-modality imaging for treatment planning

and guidance has been an area recent advancement. The vast majority of algorithms rely

on voxel-based similarity metrics (e.g. mutual information) combined with geometric-

based smoothing parameters (e.g. B-splines) (30, 31). The accuracy of these algorithms

is often sufficient when contrast is present in the images and the motion is smooth,

however, recent studies, such as the one illustrated in Figure 2(32), have indicated that

as contrast is reduced and the motion is complex and non-uniform, the accuracy reduces

substantially (33-35). In several instances (e.g. contrast-limited images, sliding interfaces)

biomechanical models have succeeded in achieving the desired level of accuracy (8, 9,

11, 17, 18, 20, 21). The successful completion of this program of research will expand

these proven models to model deformation observed between planning and intra-

procedural images for percutaneous ablation (PTA). The development of these models,

which maintain accuracy regardless of extent of contrast in the images, will enable the

safe use of deformable registration for PTA guidance (integration of pre-treatment


images) and PTA response (e.g. water loss and tissue retraction due to heating and inflammation).



Figure 2. Two methods of dose accumulation were evaluated by deforming a gel dosimeter. Morfeus was more accurate at representing the actual deformation.

#### **ELIGIBILITY**

## 1.6 Inclusion Criteria

- 1. Patients presenting with ≤ 3 liver tumors (biopsy-proven or documented by imaging) measuring 1 to 5 cm planned to undergo percutaneous thermal ablation with either microwave or radiofrequency ablation. Patients with more than 3 tumors might also be eligible in case other tumors can be treated with another curative-intended locoregional therapy (i.e. surgical resection, radiation therapy).
- 2. Ability to completely cover the target tumor with at least a 5 mm ablation margin.
- 3. Written informed consent to voluntarily participate in the study and follow-up CT scan schedule
- 4. Age > 18 years-old
- 5. Performance status 0-2 (Eastern Cooperative Oncology Group Classification [ECOG])

6. Target tumor should be visualized on contrast-enhanced CT

7. Adequate glomerular filtration rate

1.7 Exclusion Criteria

1. Active bacterial infection or fungal infection on the day of the ablation that, in the opinion

of the investigator, would interfere with safe delivery of the study procedure or with the

interpretation of study results.

2. Platelet  $< 50,000/\text{mm}^3$ .

3. INR > 1.5

4. Patients with uncorrectable coagulopathy.

5. Currently breastfeeding or pregnant (latter confirmed by serum pregnancy test).

6. Physical or psychological condition which would impair study participation.

7. ASA (American Society of Anesthesiologists) score of > 4.

8. Any other loco-regional therapies at the target lesion(s) within 30 days of the ablation

procedure.

**NUMBER OF PARTICIPANTS** 

Preliminary retrospective data on the control arm suggest that a minimum ablation margin

(MAM) of 2mm (SD 2) is generally achieved when ablation is performed without the use

of software guidance. A sample size of 50 evaluable subjects in each group will have 80%

power to detect a difference in means of -1.132 (the difference between a control arm

mean, of 2 mm and the experimental arm mean of 3.132) assuming that the common

Assuming an accrual rate of 35 patients per year, the study accrual duration will be

around 3 years, with follow-up for at least 2 years, totaling 5 years for the entire study

duration. We will have an interim look for superiority once half the evaluable subjects

(n=50) have been enrolled. A Lan-Demets spending function using an Obrien-Flemming

boundary will be used for superiority stopping boundaries. We will stop enrollment at the

control arm at our interim look if our p-value is less than 0.003. East v6.5 was used for

sample size calculation. The next 50 patients would be enrolled on the experimental arm

only to allow further development of the proposed biomechanical model on clinical

practice, as well allow other interventional radiologists at our Department to utilize it.

We plan to screen 140 subjects and expect approximately 20 subjects to be screen

failures. Furthermore, subjects after randomization who drop out due to tumor

progression, inability to clearly depict target lesions, and major complications precluding

further ablation will be considered inevaluable. To account for an expected 20%

inevaluable subjects, we will enroll a total of 120 subjects to ensure 100 evaluable

subjects.

STUDY PLAN/DESIGN

1.8 Method

RayStation® is a flexible, innovative treatment planning system. It combines

unique features like unmatched adaptive therapy capabilities, multi-criteria optimization,


optimization for HDR brachytherapy and external beam therapy with photons, electrons,

protons as well as helium and carbon ions. RayStation supports a wide range of

treatment machines, providing one control center to create biomechanical deformable

registrations using "Morfeus". Morfeus lets the investigators focus all their skill and

experience on evaluating and refining plan quality.

To investigate the impact of the proposed biomechanical model on clinical decisions during ablation guidance and end-point assessment, patients will be randomized in two

treatment arms (i.e. experimental arm - including anatomical modeling of the liver, and

control arm) with a 1:1 ratio. The primary objective is to assess whether applying

biomechanical models during percutaneous ablation will increase the minimal ablation

margins, which will be evaluated at the end of the procedure with the proposed software

on both cohorts. Additionally, two other distinct end-points will analyzed: ability of the

model to provide tumor identification for ablation probe placement on intra-procedural

non-contrast enhanced CT, and local tumor control rates achieved with the clinical

application of this model. Operating physicians will be informed in respect which arm the

patient was randomized at the time of ablation (figure 3).

Protocol No: 2019-0213 Version No: 14




Figure 3: Patient randomization flowchart

## A. Impact on tumor targeting

The clinical trial will be designed according to the optimized parameters from our retrospective analysis. The optimized biomechanical models will be used to assess the accuracy (e.g. the ability of the model to accurately describe the motion, deformation, and volume change and tumor location in the liver between the pre-ablation contrast-enhanced CT and the intra-procedural non-contrast enhanced CT) in both cohort of patients. For the control arm, no information in respect tumor location and targeting will be provided for the operating physician during ablation. Imaging processing using the biomechanical model will be performed after procedure completion. For the experimental


arm, tumor location and confirmation of appropriate targeting with ablation probe will be

performed intra-procedurally utilizing the proposed software. Differences in tumor

targeting accuracy between the two cohorts will be evaluated. If the accuracy of the cross

validation cohort is not statistically significantly different, using a paired Student's T-test

based on the preliminary retrospective results with significance defined as a p value of

less than 0.05, from the initial optimization and validation results, then the model will be

identified as complete. If the results are statistically worse, as an alternative approach,

the initial cohort of patients will be used to perform an independent optimization of the

model. Collaborations with the statistician will ensure that the appropriate power study

has been performed for the analysis. The completion of this investigation will provide the

accuracy of the present model in identifying and facilitate targeting of the liver tumors

eligible for ablation when compared to the currently utilized standard of care tumor for

tumor identification and targeting.

B. Impact on minimal ablation margins

A post ablation contrast-enhanced CT will be performed as per standard of care to

assess the minimal ablation margins. Such assessment is currently performed manually

using local rigid anatomic landmarks of the liver between the pre-ablation and post-

ablation contrast-enhanced CTs. In this aim, we will evaluate the impact on the use of the

advanced biomechanical model-based deformable alignment incorporating motion,

deformation, and ablation-related volume loss in the liver between the pre-ablation

contrast-enhanced CT and the post-ablation contrast-enhanced CT. The model will


automatically generate a minimal ablation margin on a three-dimensional Cartesian plan. Such information will be utilized by the operator physician on the experimental arm to determine whether additional ablation is needed at a particular region surrounding the target tumor using a cut-off of at  $\geq 5$  mm of minimal ablation margins in relation to the tumor borders in all planes (treatment arm). The  $\geq 5$  mm minimal ablation margin will be used to account for the margin of error of the software, which is currently 3 mm.

Frequency of total coverage of the target tumor, minimal ablation margins distance, and



Figure 4: Image fusion of pre- and post-ablation contrast-enhanced CT using the proposed biomechanical model-based deformable image registration (Morfeus). Blue line: deep learning-based segmentation of the liver; Red line: gross-tumor volume (GTV) contouring; Green line: gross-ablation volume. A minimal ablation margin of < 5 mm was detected on the latero-posterior aspect of the GTV (arrow).

need for re-ablation between the two cohorts will be analyzed to identify the impact of this model on intra-procedural decision-making.

## C. Impact on local tumor control

Rates of local recurrence following ablation in the most recent series varies from 20% to 45%. Although re-ablation on a different session is a feasible option in a minority of patients with recurrence at the ablated tumors, this incurs several disadvantages associated with the need to undergo another invasive procedure such as emotional stress, increased exposure to complications related to anesthesia and ablation procedure, radiation exposure, additional use of intravenous contrast media, and


increased associated costs. Given the complex volumetric and spatial changes of the liver post-ablation, the ability to map the previous treatment onto the new treatment plan is critical not only to avoid treatment related toxicities, but also to ensure that the patients receive adequate treatment with optimal coverage. We hypothesize that the use of this current model might improve local tumor control rates at 2-years follow-up. The completion of this aim will evaluate our hypothesis that the applied biomechanical model will improve local tumor control at 2-year when compared to the standard of care control arm.



Note: Final Analysis (n = 100 evaluable subjects)

Figure 5: Clinical Trial schema


## 1.9 Collecting Time Points

| Visit No. | Visit 1 | Visit 2 | | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 | |
|---|---|---|---|---|---|---|---|---|---|
| Visit | Screening | Ablation day | | 45 days | 3 months | 6 months | 1 year | 2 years | |
| Interval Window | Within 30 days<br>ablation | Day 0 = ablation of target lesion | | (± 14 days)<br>postablation | 3 months ( ± 1 month)<br>postablation | 6 months ( ± 1 month)<br>postablation | 12 months ( ± 1 month)<br>postablation | 24 months ( ± 3 months)<br>postablation | |
| Study Activity | | | | | | | | | |
| Informed consent | х | | | | | | | | |
| Demographic information | x | | | | | | | | |
| Medical, surgical, radiation history | soc | | | | | | | | |
| BMI and ECOG performance | soc | soc | | | soc | soc | soc | soc | soc |
| Child-Pugh, ASA scores, BCLC staging | soc | | | | SOC | soc | soc | soc | SOC |
| CBC, Coagulation, liver function, renal tests | soc | | | | SOC | soc | soc | soc | soc |
| Alpha-fetoprotein | soc | | | | SOC | soc | soc | SOC | SOC |
| Carcinoembryonic antigen | soc | | | | SOC | soc | soc | soc | soc |
| Pregnancy test | soc | | | | | | | | |
| Inclusion/exclusion | x | x | | x | | | | | |
| Concomitant medications | soc | soc | | | soc | soc | soc | SOC | soc |
| QOL questionnaire | x | | | | x | x | x | x | x |
| Numeric Pain Rating Scale | soc | | | | SOC | soc | soc | SOC | SOC |
| CT scan | soc | soc | SOC | soc | SOC | soc | soc | soc | soc |
| Ablation procedure information | | soc | soc | soc | | | | | |
| Liquid biopsy (ctDNA) | | soc | | | SOC | | soc | soc | soc |
| Physician assessment of software utility | | | | × | | | | | |
| Device user experience | | | | x | | | | | |
| Technical success assessment | | | | soc | | | | | |
| Technical efficacy assessment | | | | | soc | | | | |
| Follow-up postablation treatment | | | | | soc | soc | soc | soc | soc |

Legend: SOC: Standard of care (data collected as available per standard of care)

#### PROCEDURE TO OBTAIN CONSENT

The patients will be approached by either the Interventional Radiology Faculty or Research Staff, including research nurses and research coordinators. The principal investigator or designee who are licensed as physician in the state of Texas will obtain informed consent of participants prior to their procedure. During the consenting process patients will be educated and consented for their research participation in this study. The study will follow the Office of Research SOP04 – Informed Consent Process.

## PATIENT INFORMATION AND CONFIDENTIALITY PLAN

Confidentiality will be maintained throughout the study. An informed consent will be obtained prior to the percutaneous ablation procedure. No identifying information will


be used in any publication from this study. Patient identifiers will be available only to

the investigators for the study and will be kept in a password-protected database and

locked file cabinet. Unique patient identifiers will be used to replace patient name and

medical record number. Paper records (data forms, list of patient names and unique

identifiers), will be kept in a locked file cabinet with access granted only to study

investigators. In the conclusion of the study, patient identifiers will only be maintained

with the principal investigator to allow future review of the research. The protected

health information used in this study will not be reused, nor will it be used for other

research. As this is a prospective study, an informed consent will be obtained and

authorization to use and disclose protected health information is requested.

Morfeus, a software-aided imaging application, is located within MD Anderson

password protected behind the institutional firewall with access only granted to authorized

study investigators. Morfeus will be provided at no cost to the study participants. There

is no foreseeable injury or risk to subjects using Morfeus. Participants may withdraw from

the study at any time for any reason and are not obligated to reveal their reasons for

withdrawal, the data and test results already collected will be kept and may be used. All

study data will be stored in password-protected computers and/or locked file cabinets and

will continue to be stored securely after the study.

STATISTICAL CONSIDERATIONS

Statistical Design


The primary endpoint is to assess whether applying biomechanical models increase the minimal margins of ablated lesions properly covered by ablation on a three-dimensional analysis. The secondary endpoints of our study will compare the two arms in respect local and systemic oncological outcomes following liver ablation, procedure-related complications, and quality of life via a quality of life (QOL) questionnaire. Specifically, we will analyze the 2-years local tumor progression free-survival rates at the ablated lesions. On the experimental arm, we will evaluate the impact of software use on procedure workflow as well user's experience.

#### **Statistical Methods**

## A. Analysis Plan

Statistical analysis of this study will be the responsibility of the principal investigator (PI) and statistician. The PI and statistician will also be responsible for the appropriate conduct of an internal review for the final dataset and any study-related material to be authorized for publication.

To assess the effect of applying biomechanical image registration models during percutaneous microwave ablation, the primary endpoint of this intent-to-treat randomized trial will be on the impact of the software use on the minimal margins of ablated lesions properly covered by ablation on a three-dimensional analysis. Patients will be evenly randomized (i.e., 1:1 ratio) to two treatment arms (i.e. experimental arm - including anatomical modeling of the liver, and control arm) using the Pocock-Simon dynamic allocation method to balance the baseline covariates: tumor histology


(colorectal vs other histologies), RAS mutation (for colorectal only, yes vs. no vs.

undetermined), lesion size (<2cm, 2.0-3.0cm, >3cm-<5cm), subcapsular location,

defined as tumor within 1 cm from the liver capsule (yes vs no) and presence of multiple

lesions (yes vs. no). At the end of the study, the average minimum ablation margins will

be compared between two arms using a 2-sample t-test (or Wilcoxon rank-sum test).

The means and corresponding 95% confidence intervals will be reported for both arms

of the study.

As a secondary objective, the Kaplan-Meier method will be used to estimate local tumor progression-free survival (LTPFS) and 95% confidence intervals for the quantiles of the LTPFS function based on the method of Brookmeyer and Crowley will be calculate for each arm. Time point probabilities (e.g., 2-year LTPFS) and the associated log-log transformed pointwise 95% confidence will also be reported. A multivariate Coxproportional hazards model will be fitted to the data with ablative margin as a continuous variable to assess the significance of study arm and ablative margin size on LTPFS while simultaneously adjusting for known covariates that effect LTPFS. LTPFS will be measured from date of ablation to earliest date of progression at the ablated lesion, death. Those progression free and alive will be censored at their date of last clinic visit. Similar analysis will be used for 2-years intra-hepatic (progression at any site of the liver) progression-free survival and overall survival. Standard summary statistics will be computed for complication rates, quality of life, and liver function and compared between arms. Statistical significance will be defined as p < 0.05.


#### **B.** Randomization

A dynamic randomization method by Pocock and Simon will be used with a minimization probability parameter of 0.90. The randomization process will be controlled to ensure a balanced stratification by treatment arm for the factors listed above. Patients will be randomized to either experimental arm or no control arm using the Clinical Trial Conduct (CTC) website (https://biostatistics.mdanderson.org/ClinicalTrialConduct), which is housed on a secure server at MDACC and maintained by the MDACC Department of Biostatistics. Access to the website will be gained through usernames and passwords provided by the MDACC Department of Biostatistics to the clinical team. Training on the use of the CTC website to randomize patients on the study will be provided by the biostatistical collaborators. This is an open-label trial with stratified randomization. When a patient is enrolled on the study, the research nurse or coordinator of the study will enter patient's information including medical record number and stratification factors. Through the web interface, after the randomization button is clicked, the result of the randomization will be displayed on the screen for users to view. All data on randomization will be stored in a secure SQL server database.

## PROTOCOL MONITORING PLAN

MD Anderson's Data Safety Monitoring Board (DSMB) will monitor the conduct of the study. The principal investigator will be responsible for the management of the protocol. Identifiers (name, medical record number) will be collected but will be replaced by study numbers in the analytical file. They key linking these numbers will be retained in a locked file by the principal investigator. All study personnel have


completed training in methods of maintaining the confidentiality of health information.

Electronic records will be stored on password protected institution computers behind the institution firewall. Only the principal investigator and research staff in Interventional Radiology will have access to the study. Data will not be transferred to laptop computers that are removed from the institution. Complete confidentiality will be maintained during this evaluation, manuscript preparation and submission. Information from individual Case Report Forms (CRFs) will be saved in an institutionally-based and approved electronic database. Adverse events such as inaccurate tumor localization and ablation coverage, as well as subsequent local tumor progression will be captured and recorded in OnCore.

#### **DATA COLLECTION PLAN**

All subjects will be registered in OnCore and data will be entered in an UT MD Anderson Cancer Center approved electronic database. The institutionally approved database is a secure, web-based application with controlled access designed to support data capture for research studies, providing: 1) an intuitive interface for validated data entry; 2) audit trails for tracking data manipulation and export procedures; 3) automated export procedures for seamless downloads to common statistical packages; and 4) procedures for importing data from external sources. It is hosted on a secure server by MD Anderson Cancer Center that has undergone an annual Governance Risk & Compliance Assessment by MD Anderson's Information Security Office and found to be compliant with HIPAA, Texas Administrative Codes 202-203, University of Texas Policy


165, federal regulations outlined in 21CFR Part 11, and UTMDACC Institutional Policy #ADM0335.

Those having access to the data include the study PI and research team personnel. Users are authenticated against MDACC's Active Directory system. The application is accessed through Secure Socket Layer (SSL). All personal identifying information will be removed from the data when it is exported for analysis.

Following publication, study data will be archived in the electronic database indefinitely, since study data may be useful for future research studies performed under separate IRB approved protocols. Since this is a secure electronic database with controlled access, and because subject identifiers may be needed to link study data to data from other sources under future IRB approved protocols, subject identifying information will be retained in the archived database. No specific subject identifiers will be collected in this study. We acknowledge that there is a theoretical chance that the participants may be identified from their combined responses to the demographic questions. However, no attempt will be made by the research personnel to identify the survey respondents. Also, data will only be reported in aggregate form. The demographic information in the survey, along with all other survey responses, will be stored securely in the database. Up to five fully deidentified CT images will be shared with RaySearch Laboratories for joint development purposes directly related to the NIH-funded Academic-Industry Partnership R01 for the COVER-ALL clinical trial and project. RaySearch Laboratories is the industry partner for this grant.


#### REFERENCES

- 1. Bruix J, Reig M, Sherman M. Evidence-Based Diagnosis, Staging, and Treatment of Patients With Hepatocellular Carcinoma. Gastroenterology. 2016;150(4):835-53.
- 2. Abdalla EK, Vauthey JN, Ellis LM, Ellis V, Pollock R, Broglio KR, et al. Recurrence and outcomes following hepatic resection, radiofrequency ablation, and combined resection/ablation for colorectal liver metastases. Ann Surg. 2004;239(6):818-25; discussion 25-7.
- 3. Van Cutsem E, Cervantes A, Adam R, Sobrero A, Van Krieken JH, Aderka D, et al. ESMO consensus guidelines for the management of patients with metastatic colorectal cancer. Ann Oncol. 2016;27(8):1386-422.
- 4. Ruers T, Van Coevorden F, Punt CJ, Pierie JE, Borel-Rinkes I, Ledermann JA, et al. Local Treatment of Unresectable Colorectal Liver Metastases: Results of a Randomized Phase II Trial. J Natl Cancer Inst. 2017;109(9).
- 5. Solbiati L, Ahmed M, Cova L, Ierace T, Brioschi M, Goldberg SN. Small liver colorectal metastases treated with percutaneous radiofrequency ablation: local response rate and long-term survival with up to 10-year follow-up. Radiology. 2012;265(3):958-68.
- 6. Benson AB, 3rd, Bekaii-Saab T, Chan E, Chen YJ, Choti MA, Cooper HS, et al. Metastatic colon cancer, version 3.2013: featured updates to the NCCN Guidelines. J Natl Compr Canc Netw. 2013;11(2):141-52; quiz 52.
- 7. Shady W, Petre EN, Gonen M, Erinjeri JP, Brown KT, Covey AM, et al. Percutaneous Radiofrequency Ablation of Colorectal Cancer Liver Metastases: Factors Affecting Outcomes--A 10-year Experience at a Single Center. Radiology. 2016;278(2):601-11.
- 8. Al-Mayah A, Moseley J, Brock KK. Contact surface and material nonlinearity modeling of human lungs. Phys Med Biol. 2008;53(1):305-17.
- 9. Al-Mayah A, Moseley J, Hunter S, Velec M, Chau L, Breen S, et al. Biomechanical-based image registration for head and neck radiation treatment. Phys Med Biol. 2010;55(21):6491-500.
- 10. Al-Mayah A, Moseley J, Velec M, Brock K. Toward efficient biomechanical-based deformable image registration of lungs for image-guided radiotherapy. Phys Med Biol. 2011;56(15):4701-13.
- 11. Al-Mayah A, Moseley J, Velec M, Brock KK. Sliding characteristic and material compressibility of human lung: parametric study and verification. Med Phys. 2009;36(10):4625-33.
- 12. Al-Mayah A, Moseley J, Velec M, Hunter S, Brock K. Deformable image registration of heterogeneous human lung incorporating the bronchial tree. Med Phys. 2010;37(9):4560-71.

Protocol No: 2019-0213 Version No: 14


13. Alonzo-Proulx O, Packard N, Boone JM, Al-Mayah A, Brock KK, Shen SZ, et al. Validation of a method for measuring the volumetric breast density from digital mammograms. Phys Med Biol. 2010;55(11):3027-44.

- 14. Breen SL, Publicover J, De Silva S, Pond G, Brock K, O'Sullivan B, et al. Intraobserver and interobserver variability in GTV delineation on FDG-PET-CT images of head and neck cancers. Int J Radiat Oncol Biol Phys. 2007;68(3):763-70.
- 15. Brierley JD, Dawson LA, Sampson E, Bayley A, Scott S, Moseley JL, et al. Rectal motion in patients receiving preoperative radiotherapy for carcinoma of the rectum. Int J Radiat Oncol Biol Phys. 2011;80(1):97-102.
- 16. Brock KK, Dawson LA, Sharpe MB, Moseley DJ, Jaffray DA. Feasibility of a novel deformable image registration technique to facilitate classification, targeting, and monitoring of tumor and normal tissue. Int J Radiat Oncol Biol Phys. 2006;64(4):1245-54.
- 17. Brock KK, Hawkins M, Eccles C, Moseley JL, Moseley DJ, Jaffray DA, et al. Improving image-guided target localization through deformable registration. Acta Oncol. 2008;47(7):1279-85.
- 18. Brock KK, Nichol AM, Menard C, Moseley JL, Warde PR, Catton CN, et al. Accuracy and sensitivity of finite element model-based deformable registration of the prostate. Med Phys. 2008;35(9):4019-25.
- 19. Brock KK, Sharpe MB, Dawson LA, Kim SM, Jaffray DA. Accuracy of finite element model-based multi-organ deformable image registration. Med Phys. 2005;32(6):1647-59.
- 20. Eccles C, Brock KK, Bissonnette JP, Hawkins M, Dawson LA. Reproducibility of liver position using active breathing coordinator for liver cancer radiotherapy. Int J Radiat Oncol Biol Phys. 2006;64(3):751-9.
- 21. Eccles CL, Dawson LA, Moseley JL, Brock KK. Interfraction liver shape variability and impact on GTV position during liver stereotactic radiotherapy using abdominal compression. Int J Radiat Oncol Biol Phys. 2011;80(3):938-46.
- 22. Hawkins MA, Brock KK, Eccles C, Moseley D, Jaffray D, Dawson LA. Assessment of residual error in liver position using kV cone-beam computed tomography for liver cancer high-precision radiation therapy. Int J Radiat Oncol Biol Phys. 2006;66(2):610-9.
- 23. Kirilova A, Lockwood G, Choi P, Bana N, Haider MA, Brock KK, et al. Three-dimensional motion of liver tumors using cine-magnetic resonance imaging. Int J Radiat Oncol Biol Phys. 2008;71(4):1189-95.
- 24. Nguyen TN, Moseley JL, Dawson LA, Jaffray DA, Brock KK. Adapting population liver motion models for individualized online image-guided therapy. Conf Proc IEEE Eng Med Biol Soc. 2008;2008:3945-8.
- 25. Niu CJ, Foltz WD, Velec M, Moseley JL, Al-Mayah A, Brock KK. A novel technique to enable experimental validation of deformable dose accumulation. Med Phys. 2012;39(2):765-76.
- 26. Velec M, Moseley JL, Craig T, Dawson LA, Brock KK. Accumulated dose in liver stereotactic body radiotherapy: positioning, breathing, and deformation effects. Int J Radiat Oncol Biol Phys. 2012;83(4):1132-40.

Protocol No: 2019-0213 Version No: 14


27. Velec M, Moseley JL, Eccles CL, Craig T, Sharpe MB, Dawson LA, et al. Effect of breathing motion on radiotherapy dose accumulation in the abdomen using deformable registration. Int J Radiat Oncol Biol Phys. 2011;80(1):265-72.

- 28. Voroney JP, Brock KK, Eccles C, Haider M, Dawson LA. Prospective comparison of computed tomography and magnetic resonance imaging for liver cancer delineation using deformable image registration. Int J Radiat Oncol Biol Phys. 2006;66(3):780-91.
- 29. White EA, Brock KK, Jaffray DA, Catton CN. Inter-observer variability of prostate delineation on cone beam computerised tomography images. Clin Oncol (R Coll Radiol). 2009;21(1):32-8.
- 30. Brock KK, Deformable Registration Accuracy C. Results of a multi-institution deformable registration accuracy study (MIDRAS). Int J Radiat Oncol Biol Phys. 2010;76(2):583-96.
- 31. Kashani R, Hub M, Balter JM, Kessler ML, Dong L, Zhang L, et al. Objective assessment of deformable image registration in radiotherapy: a multi-institution study. Med Phys. 2008;35(12):5944-53.
- 32. Velec M, Juang T, Moseley JL, Oldham M, Brock KK. Utility and validation of biomechanical deformable image registration in low-contrast images. Pract Radiat Oncol. 2015;5(4):e401-8.
- 33. Kirby N, Chuang C, Pouliot J. A two-dimensional deformable phantom for quantitatively verifying deformation algorithms. Med Phys. 2011;38(8):4583-6.
- 34. Kirby N, Chuang C, Ueda U, Pouliot J. The need for application-based adaptation of deformable image registration. Med Phys. 2013;40(1):011702.
- 35. Nie K, Chuang C, Kirby N, Braunstein S, Pouliot J. Site-specific deformable imaging registration algorithm selection using patient-based simulated deformations. Med Phys. 2013;40(4):041911.


# **QUESTIONNAIRES**

# Software user's experience

| Specific Use | Definition | Software helped me<br>(1: no; 2: somewhat;<br>3: yes) | Comments |
|---|---|---|---|
| Probe Placement | Ability to understand probe positioning in relation to the target lesion | | |
| Ablation confirmation | Evaluating technical success of the procedure (full coverage of the tumor) | | |


# **Procedure Details**

| Variable measured | Definition | Answer |
|--------------------------------|-------------------|--------|
| Number of probes | 1 – 3 | |
| utilized on the target lesions | 1-3 | |
| Number of | 0-3 | |
| overlapping ablations | | |
| Total duration of | la miauta (F. 20) | |
| ablation (counting overlaps) | In minutes (5-20) | |
| Post-ablation | | |
| Contrast-enhanced | Yes/No | |
| CT after first round of | | |
| ablation? | , | |
| Need to re-ablation? | Yes / no | |
| Number of probes | _ | |
| utilized on the target | 1-3 | |
| lesions | | |
| Number of | 0-3 | |
| overlapping ablations | | |
| Total duration of | L'. L. (F. 20) | |
| ablation (counting overlaps) | In minutes (5-20) | |
| Post-ablation | | |
| Contrast-enhanced | | |
| CT after second | Yes/No | |
| round of ablation? | | |
| Need to re-ablation? | Yes / no | |
| Number of probes | | |
| utilized on the target | 1-3 | |
| lesions | | |
| Number of | 0-3 | |
| overlapping ablations | 0-3 | |
| Total duration of | | |
| ablation (counting | In minutes (5-20) | |
| overlaps) | | |

Protocol No: 2019-0213 Version No: 14


## **QUALITY OF LIFE QUESTTIONAIRE**

## **EORTC QLQ-C30 Questionnaire**

We are interested in some things about you and your health. Please answer all of the questions yourself by circling the number that best applies to you. There are no "right" or "wrong" answers.

| | | Not at<br>All | A<br>Little | Quite<br>a Bit | Very<br>Much |
|---|---|---|---|---|---|
| | o you have any trouble doing strenuous activities,<br>ke carrying a heavy shopping bag or a suitcase? | 1 | 2 | 3 | 4 |
| 2. D | o you have any trouble taking a <u>long</u> walk? | 1 | 2 | 3 | 4 |
| | o you have any trouble taking a <u>short</u> walk outside of the ouse? | 1 | 2 | 3 | 4 |
| 4. D | o you need to stay in bed or a chair during the day? | 1 | 2 | 3 | 4 |
| | o you need help with eating, dressing, washing<br>ourself or using the toilet? | 1 | 2 | 3 | 4 |
| During the past week: | | Not at<br>All | A<br>Little | Quite<br>a Bit | Very<br>Much |
| | Vere you limited in doing either your work or other daily ctivities? | 1 | 2 | 3 | 4 |
| | Vere you limited in pursuing your hobbies pr<br>ther leisure time activities? | 1 | 2 | 3 | 4 |
| 8. W | Vere you short of breath? | 1 | 2 | 3 | 4 |
| 9. H | lave you had pain? | 1 | 2 | 3 | 4 |
| 10. D | oid you need to rest? | 1 | 2 | 3 | 4 |
| 11. H | lave you had trouble sleeping? | 1 | 2 | 3 | 4 |
| 12. H | lave you felt weak? | 1 | 2 | 3 | 4 |
| 13. H | lave you lacked appetite? | 1 | 2 | 3 | 4 |
| 14. H | lave you felt nauseated? | 1 | 2 | 3 | 4 |
| 15. H | lave you vomited? | 1 | 2 | 3 | 4 |
| 16. H | lave you been constipated? | 1 | 2 | 3 | 4 |


